CLINICAL TRIAL: NCT01128621
Title: A Study in Type 2 Diabetic Subjects on Stable Metformin Therapy to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Co-administering Single and Multiple Oral Doses of GSK1292263
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 113132
Record Dates: First submitted 2010-02-12; First posted 2010-05-24 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Pharmacokinetics; Glucose; Safety; Male; Female; Metformin; Pharmacodynamics; Tolerability; Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (1-(3-isopropyl-1,2,4-oxadiazol-5-yl)piperidin-4-yl)methyl methanesulfonate; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A (Other): Part A is open label, in T2DM subjects on established metformin monotherapy. Subjects will receive a single dose of GSK1292263 with food. This will permit a comparison of GSK1292263 exposures in this cohort with those observed in study GPR111598 in which T2DM subjects were drug naïve or washed off prior anti-diabetic medications.
  Interventions: Drug: GSK1292263
- Part B - PLA (Placebo Comparator): Part B is a single-blind, randomized, placebo-controlled, 4-arm cohort of 48 subjects dosed for 14 days with one of two doses of GSK1292263 BID, placebo BID or open-label sitagliptin 50mg BID. It is being conducted to assess safety, tolerability, PK and PD of GSK1292263 and open-label sitagliptin after 14-days of dosing in T2DM subjects already taking metformin monotherapy.
  Interventions: Drug: GSK1292263 matching placebo
- Part B - Active (Active Comparator): Part B is a single-blind, randomized, placebo-controlled, 4-arm cohort of 48 subjects dosed for 14 days with one of two doses of GSK1292263 BID, placebo BID or open-label sitagliptin 50mg BID. It is being conducted to assess safety, tolerability, PK and PD of GSK1292263 and open-label sitagliptin after 14-days of dosing in T2DM subjects already taking metformin monotherapy.
  Interventions: Drug: GSK1292263
- Part B - Sitagliptin (Active Comparator): Part B is a single-blind, randomized, placebo-controlled, 4-arm cohort of 48 subjects dosed for 14 days with one of two doses of GSK1292263 BID, placebo BID or open-label sitagliptin 50mg BID. It is being conducted to assess safety, tolerability, PK and PD of GSK1292263 and open-label sitagliptin after 14-days of dosing in T2DM subjects already taking metformin monotherapy.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: GSK1292263 — Tablet
  Arms: Part A; Part B - Active
Drug: GSK1292263 matching placebo — Tablet
  Arms: Part B - PLA
Drug: Sitagliptin — Tablet
  Arms: Part B - Sitagliptin

SUMMARY:
A study in type 2 diabetic subjects on stable metformin therapy to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of co-administering single and multiple oral doses of GSK1292263

DETAILED DESCRIPTION:
This study will investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of GSK1292263 when co-administered with metformin. The study will be in 2 parts. Part A will determine the PK of GSK1292263 following single day dosing of type 2 diabetes (T2DM) subjects on metformin. Part B will investigate the effects of 14d of co-dosing of GSK1292263 BID, 50mg BID of sitagliptin or placebo to 48 T2DM subjects taking metformin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 - 65 years of age, inclusive.
* Females of non-childbearing potential.
* Male subjects willing to employ appropriate contraception.
* Except as noted elsewhere, subjects should have no significant known medical conditions other than T2DM that would affect the safety of the subject or the objectives of the study.
* BMI (body mass index) within the range 21.8-37.5 kg/m2.
* T2DM diagnosed by American Diabetes Association criteria for at least 3 month prior to screening.
* Currently on stable metformin therapy.
* Fasting plasma glucose <= 250mg/dL.
* HbA1c between 6.5 and 11.0%.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with right bundle branch block. Subjects with left bundle branch block are not eligible.
* AST and ALT < 2xULN; alkaline phosphatase and bilirubin <=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). Subjects with Gilbert's syndrome are allowed to participate in the study.

Exclusion Criteria:

* Positive for Hepatitis B or C, or HIV.
* History of uncorrected thyroid dysfunction or an abnormal thyroid function test.
* History of ketoacidosis or lactic acidosis.
* Fasting triglycerides > 450mg/dL.
* For females a hemoglobin < 11.5g/dL, and for males a hemoglobin < 12.5g/dL.
* Positive drug/alcohol screen.
* Smoking.
* If female is pregnant or has a positive pregnancy test or is lactating.
* Significant renal disease.
* Significant ECG abnormalities.
* Systolic blood pressure > 150mmHg or <80mmHg or diastolic blood pressure > 95mmHg or <60mmHg at screening.
* Previous use of insulin as a treatment within 3 months of screening, or for >2 weeks when used for acute illness in the last 12 months prior to screening, or if used for more than 1 year when associated with gestational diabetes mellitus.
* History of: clinically significant symptoms of gastroparesis; symptomatic cholelithiasis or obstructive or inflammatory gallbladder disease within 3 months prior to screening; gastrointestinal disease that could affect fat or bile acid absorption, or the pharmacokinetics or pharmacodynamics of the study drugs, including inflammatory bowel disease, chronic diarrhea, Crohn's or malabsorption syndromes within the past year; gastrointestinal surgery that may affect the pharmacokinetics or pharmacodynamics of the study drugs; or, chronic or acute pancreatitis.
* History of regular alcohol consumption within 6 months.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months.
* Has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Is taking prohibited medications. In Parts A and B, subjects will not be allowed to wash-off of unapproved anti-diabetic medications in order to qualify for participation in this study. • Subjects must wash out from the following medications during the 7-day period prior to first dose, and must remain off these medications through discharge on Day 2 (Part A) or Day 15 (Part B): all statin agents, fat absorption blocking agents, bile acid sequestrants. Fibrates must be washed out for a 14-day period prior to first dose. • Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Unwilling to abstain from: Caffeine-or xanthine-containing products from Day -7 until D2 (Part A) or Day -7 through Day 15 (Part B); use of illicit drugs or nicotine-containing products; alcohol from Day -7 prior to dosing until D2 (Part A) or Day -7 through Day 15 (Part B); Consumption of red wine, Seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication until collection of the final pharmacokinetic blood samples.
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation. This includes sensitivity to heparin or heparin-induced thrombocytopenia, if heparin will be used to maintain catheter patency.
* Where participation in the study would result in donation of blood in excess of approximately 500mL within a 56 day period.
* Subject is either an immediate family member of a participating investigator, study coordinator, employee of an investigator; or is a member of the staff conducting the study.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-11-23 (Actual); Primary Completion 2010-04-12 (Actual); Study Completion 2010-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Miami, Florida

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Nunez DJ, Bush MA, Collins DA, McMullen SL, Gillmor D, Apseloff G, Atiee G, Corsino L, Morrow L, Feldman PL. Gut hormone pharmacology of a novel GPR119 agonist (GSK1292263), metformin, and sitagliptin in type 2 diabetes mellitus: results from two randomized studies. PLoS One. 2014 Apr 3;9(4):e92494. doi: 10.1371/journal.pone.0092494. eCollection 2014. PMID 24699248
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113132 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at two study centers in the United States from 23 November 2009 up to 12 April 2010. The study consisted of open label Part A and single-blind Part B. Total 6 participants were randomized in Part A whereas total 67 participants were randomized in Part B.
Groups:
- Part A: GSK1292263 300 mg: Participants received a single dose of oral 300 milligrams (mg) tablet of GSK1292263 on Day 1 immediately after eating the breakfast meal. Participants also received their usual metformin monotherapy (>=1000 mg per day).
- Part B: GSK1292263 75 mg/300 mg/ 600 mg: Participants received one of three dosing regimens of GSK1292263: 75 mg twice daily (BID) (as 1 x 75 mg tablet GSK1292263 + 2 placebo tablets in morning and evening), 300 mg BID (as 1 x 200 mg tablet + 1 x 75 mg tablet + 1 x 25 mg tablet GSK1292263 in morning and evening) and 600 mg once daily (QD) (as 3 x 200 mg tablets GSK1292263 in morning + 3 x placebo tablets in evening) or matching placebo BID (as 3 x placebo tablets in morning and evening), or open-label sitagliptin 50 mg BID for 14 days. Seven days before enrollment in Part B, participants taking metformin three times daily (TID) or using an extended-release formulation were converted to the equivalent total daily dose of immediate release metformin administered BID.
Period: Part A: GSK1292263 300 mg
Arm/Group | Part A: GSK1292263 300 mg | Part B: GSK1292263 75 mg/300 mg/ 600 mg
Started | 6 | 0
Completed | 6 | 0
Not Completed | 0 | 0
Period: Part B: GSK1292263 75 mg/300 mg/ 600 mg
Arm/Group | Part A: GSK1292263 300 mg | Part B: GSK1292263 75 mg/300 mg/ 600 mg
Started | 0 | 67
Completed | 0 | 65
Not Completed | 0 | 2
Not completed — Reached defined stopping criteria | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Part A: GSK1292263 300 mg: Participants received a single dose of oral 300 mg tablet of GSK1292263 on Day 1 immediately after eating the breakfast meal. Participants also received their usual metformin monotherapy (>=1000 mg per day).
- Total: Total of all reporting groups
Arm/Group | Part A: GSK1292263 300 mg | Part B: GSK1292263 75 mg/300 mg/ 600 mg | Total
Number analyzed (Participants) | 6 | 67 | 73
Age, Customized [Count of Participants; unit: Participants]
  36 to 65 Years | 6 | 67 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 28 | 29
  Male | 5 | 39 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 4 | 61 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs) (Part A)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury.
Time Frame: Up to 10 days after discharge (Day 2) in Part A
Population: Safety Population consisted of all participants enrolled in the study and who had received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Participants received a single dose of oral 300 mg tablet of GSK1292263 on Day 1 immediately after eating the breakfast meal. Participants also received their usual metformin monotherapy (>=1000 mg per day).
Arm/Group | Part A
Number analyzed (Participants) | 6
Participants
  Any AE | 0
  Any SAE | 0

2. Primary Outcome: Number of Participants With Any AEs and Serious Adverse Events SAEs (Part B)
Description: as for outcome 1
Time Frame: Up to 10 days after discharge (Day 15) in Part B
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received 3 tablets of matching placebo BID along with metformin for 14 days
- GSK1292263 75 mg: Participant received 1 tablet of 75 mg of GSK1292263 and 2 tablets of matching placebo along with metformin BID for 14 days
- GSK1292263 300 mg: Participant received 1 tablet of 200 mg, 1 tablet of 75 mg and 1 tablet of 25 mg (all GSK1292263) along with metformin BID for 14 days
- GSK1292263 600 mg: Participant received 3 tablet of 200 mg of GSK1292263 in the morning and 3 tablets of matching placebo in the evening along with metformin for 14 days.
- Sitagliptin 50 mg: Participant received 50 mg of Sitagliptin BID along with metformin for 14 days.
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 15 | 13
Participants
  Any AE | 2 | 3 | 3 | 4 | 5
  Any SAE | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Hematology Values of Potential Clinical Importance (PCI) (Part A)
Description: Blood samples for hematology assessments were collected at screening, fasting (Day -1), at 24hr post- dose (morning of Day 2), and at follow-up. Hematology parameter: Total Neutrophil count was assessed for abnormal value of PCI. The range of PCI value was: <0.83 x lower limit normal (LLN) with unit x10^9 per liter
Time Frame: Up to 10 days after discharge (Day 2) in Part A
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 6
Participants | 1

4. Primary Outcome: Number of Participants With Abnormal Hematology Values of PCI (Part B)
Description: Blood samples for hematology assessments were collected at screening, on Day -2 (non-fasting), and prior to breakfast (early in the morning, fasting) on Days 1, 7, and on Day 15 prior to checkout, (=24hrs post-dose), and at follow-up. Hematology parameters: Hematocrit (unit: ratio) and hemoglobin (unit: grams per liter [g/L]), were assessed for abnormal values of PCI. The PCI range for hematocrit was: >0.075 decrease from Baseline (low), >1.02 x upper limit normal (ULN) (high-male), >1.17 x ULN (high-female). The PCI range for hemoglobin was: >25 decrease from Baseline (low), >1.03 x ULN (high-male), >1.13 x ULN (high-female). Data has been presented for the number of participants with hematology data values high from the PCI range in a consolidated format.
Time Frame: Up to 10 days after discharge (Day 15) in Part B
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Sitagliptin 50mg: Participant received 50 mg of Sitagliptin BID along with metformin for 14 days.
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50mg
Number analyzed (Participants) | 14 | 13 | 12 | 15 | 13
Participants
  Hematocrit, high | 0 | 1 | 0 | 1 | 0
  Hemoglobin, high | 0 | 1 | 1 | 1 | 1

5. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Values of PCI (Part A)
Description: Blood samples for chemistry assessments were collected at screening, fasting (Day -1), at 24hr post- dose (morning of Day 2), and at follow-up.
  Clinical chemistry parameter: Glucose (unit: millimoles per liter [mmol/L]) was assessed for abnormal high value of PCI. The normal range was 3.6 to 5.5 mmol/L
Time Frame: Up to 10 days after discharge (Day 2) in Part A
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 6
Participants | 1

6. Primary Outcome: Number of Participants With Abnormal Clinical Chemistry Values of PCI (Part B)
Description: Blood samples for chemistry assessments were collected at screening, on Day -2 (non-fasting), and prior to breakfast (early in the morning, fasting) on Days 1, 7, and on Day 15 prior to checkout, (=24hrs post-dose), and at follow-up. Clinical chemistry parameters: Aspartate amino transferase (unit: international unit per liter [IU/L]) and Total bilirubin (unit: micromoles per liter (µmol/L) were assessed for abnormal values of PCI. For aspartate aminotransferase the PCI range was >=2 x ULN (high). For total bilirubin the PCI range was >=1.5 x ULN (high).
Time Frame: Up to 10 days after discharge (Day 15) in Part B
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 15 | 13
Participants
  Aspartate aminotransferase, high | 0 | 0 | 0 | 1 | 0
  Total bilirubin, high | 0 | 0 | 0 | 0 | 1

7. Primary Outcome: Number of Participants With Abnormal Urinalysis Data Values by Dipstick Method (Part A)
Description: Urinalysis parameters: Urine occult blood, Urine Glucose, Urine ketones and Urine protein were assessed for abnormal findings by dipstick analysis. The abnormalities were presented as trace, 1+, 2+ and 3+. Trace indicates lowest concentration of the mentioned parameters in urine and 3+ indicates highest concentration. Concentration of 3+ indicates worse outcome.
Time Frame: Up to 10 days after discharge (Day 2) in Part A
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 6
Participants
  Urine occult blood, Day 1, 24 hours, trace | 1
  Urine occult blood, follow up, trace | 1
  Urine glucose, Day 1, 24 hours, 3+ | 1
  Urine glucose, follow up, 3+ | 1
  Urine glucose, follow up, trace | 2
  Urine ketones, follow up, trace | 2
  Urine protein, Day 1, 24 hours, trace | 1
  Urine protein, follow up, trace | 2

8. Primary Outcome: Number of Participants With Abnormal Urinalysis Data Values (Part B)
Description: Urinalysis parameters: Urine occult blood, Urine glucose, Urine ketones, Urine protein, White blood cells were assessed for abnormal findings by dipstick analysis. The abnormal findings were presented as trace, 1+, 2+ and 3+. Trace indicates lowest concentration of the mentioned parameters in urine and 3+ indicates highest concentration. Concentration of 3+ indicates worse outcome.
Time Frame: Up to 10 days after discharge (Day 15) in Part B
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 15 | 13
Participants
  Urine occult blood, Day 1, pre-breakfast, 3+ | 0 | 0 | 0 | 0 | 1
  Urine occult blood, Day 1, pre-breakfast, trace | 1 | 2 | 0 | 0 | 0
  Urine occult blood, Day 7, pre-breakfast, trace | 1 | 1 | 1 | 0 | 0
  Urine occult blood, Day 14, 24 hours, trace: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Urine occult blood, Day 14, 24 hours, trace | 2 | 2 | 0 | 2 | 0
  Urine occult blood, follow up, trace: number analyzed (Participants) | 13 | 10 | 12 | 12 | 12
  Urine occult blood, follow up, trace | 0 | 2 | 0 | 1 | 0
  Urine glucose, Day 1, pre-breakfast, 1+ | 1 | 0 | 0 | 0 | 0
  Urine glucose, Day 1, pre-breakfast, 2+ | 1 | 0 | 0 | 0 | 0
  Urine glucose, Day 1, pre-breakfast, 3+ | 1 | 0 | 1 | 1 | 0
  Urine glucose, Day 1, pre-breakfast, trace | 0 | 2 | 0 | 1 | 1
  Urine glucose, Day 7, pre-breakfast, 1+ | 1 | 0 | 0 | 0 | 0
  Urine glucose, Day 7, pre-breakfast, 2+ | 0 | 0 | 0 | 1 | 0
  Urine glucose, Day 7, pre-breakfast, trace | 1 | 0 | 2 | 0 | 0
  Urine glucose, Day 14, 24 hours, 3+: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Urine glucose, Day 14, 24 hours, 3+ | 0 | 0 | 1 | 1 | 0
  Urine glucose, Day 14, 24 hours, trace: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Urine glucose, Day 14, 24 hours, trace | 0 | 1 | 1 | 1 | 0
  Urine glucose, follow up, 1+: number analyzed (Participants) | 13 | 12 | 12 | 13 | 12
  Urine glucose, follow up, 1+ | 0 | 0 | 1 | 0 | 0
  Urine glucose, follow up, 2+: number analyzed (Participants) | 13 | 12 | 12 | 13 | 12
  Urine glucose, follow up, 2+ | 1 | 2 | 0 | 0 | 0
  Urine glucose, follow up, 3+: number analyzed (Participants) | 13 | 12 | 12 | 13 | 12
  Urine glucose, follow up, 3+ | 1 | 0 | 4 | 2 | 0
  Urine glucose, follow up, trace: number analyzed (Participants) | 13 | 12 | 12 | 13 | 12
  Urine glucose, follow up, trace | 2 | 2 | 1 | 2 | 1
  Urine ketones, Day 1, pre-breakfast, trace | 0 | 1 | 0 | 1 | 0
  Urine ketones, Day 7, pre-breakfast, trace | 0 | 0 | 1 | 2 | 0
  Urine ketones, Day 14, 24 hours, trace: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Urine ketones, Day 14, 24 hours, trace | 0 | 1 | 2 | 0 | 0
  Urine ketones, follow up, 1+: number analyzed (Participants) | 13 | 12 | 12 | 13 | 12
  Urine ketones, follow up, 1+ | 0 | 0 | 1 | 0 | 0
  Urine ketones, follow up, trace: number analyzed (Participants) | 13 | 12 | 12 | 13 | 12
  Urine ketones, follow up, trace | 0 | 0 | 1 | 4 | 0
  Urine protein, Day 1, pre-breakfast, trace | 0 | 2 | 0 | 2 | 1
  Urine protein, Day 7, pre-breakfast, 1+ | 0 | 0 | 0 | 1 | 0
  Urine protein, Day 7, pre-breakfast, trace | 1 | 2 | 1 | 1 | 0
  Urine protein, Day 14, 24 hours, trace: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Urine protein, Day 14, 24 hours, trace | 0 | 2 | 3 | 1 | 0
  Urine protein, follow up, 1+: number analyzed (Participants) | 13 | 12 | 12 | 13 | 12
  Urine protein, follow up, 1+ | 1 | 1 | 0 | 0 | 0
  Urine protein, follow up, 2+: number analyzed (Participants) | 13 | 12 | 12 | 13 | 12
  Urine protein, follow up, 2+ | 1 | 0 | 1 | 0 | 0
  Urine protein, follow up, trace: number analyzed (Participants) | 13 | 12 | 12 | 13 | 12
  Urine protein, follow up, trace | 3 | 3 | 4 | 4 | 1
  White blood cells, Day 1, pre-breakfast, 1+: number analyzed (Participants) | 13 | 11 | 10 | 9 | 11
  White blood cells, Day 1, pre-breakfast, 1+ | 2 | 1 | 2 | 0 | 0
  White blood cells, Day 1, pre-breakfast, trace: number analyzed (Participants) | 13 | 11 | 10 | 9 | 11
  White blood cells, Day 1, pre-breakfast, trace | 2 | 1 | 1 | 1 | 1
  White blood cells, Day 7, pre-breakfast, 1+: number analyzed (Participants) | 13 | 11 | 10 | 9 | 11
  White blood cells, Day 7, pre-breakfast, 1+ | 0 | 0 | 1 | 0 | 0
  White blood cells, Day 7, pre-breakfast, trace: number analyzed (Participants) | 13 | 11 | 10 | 9 | 11
  White blood cells, Day 7, pre-breakfast, trace | 1 | 1 | 2 | 0 | 1
  White blood cells, Day 14, 24 hours, 1+: number analyzed (Participants) | 13 | 11 | 10 | 9 | 11
  White blood cells, Day 14, 24 hours, 1+ | 0 | 1 | 0 | 0 | 1
  White blood cells, Day 14, 24 hours, trace: number analyzed (Participants) | 13 | 11 | 10 | 9 | 11
  White blood cells, Day 14, 24 hours, trace | 5 | 1 | 0 | 1 | 1
  White blood cells, follow up, 1+: number analyzed (Participants) | 12 | 10 | 10 | 7 | 10
  White blood cells, follow up, 1+ | 0 | 1 | 0 | 0 | 0
  White blood cells, follow up, 2+: number analyzed (Participants) | 12 | 10 | 10 | 7 | 10
  White blood cells, follow up, 2+ | 1 | 0 | 0 | 0 | 0
  White blood cells, follow up, trace: number analyzed (Participants) | 12 | 10 | 10 | 7 | 10
  White blood cells, follow up, trace | 2 | 0 | 1 | 0 | 0

9. Primary Outcome: Mean Value of Urine Albumin at Follow up (Part A)
Description: Urine samples were collected at screening, Day -1, at 24hr post- dose (Day 2), and at follow-up. Urine albumin was assessed using quantitative analysis.
Time Frame: Up to 10 days after discharge (Day 2) in Part A
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: milligrams per liter (mg/L)
Groups:
- Arm A: Participants received a single dose of oral 300 mg tablet of GSK1292263 on Day 1 immediately after eating the breakfast meal. Participants also received their usual metformin monotherapy (>=1000 mg per day).
Arm/Group | Arm A
Number analyzed (Participants) | 1
milligrams per liter (mg/L) | 6.0 (NA) — Not available as only 1 participant was analyzed

10. Primary Outcome: Mean Value of Urine Albumin (Part B)
Description: Urine samples were collected at screening, on Day -2, and on Days 1, 7, 15 and at follow-up. Urine albumin was assessed using quantitative analysis.
Time Frame: Up to 10 days after discharge (Day 15) in Part B
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 15 | 13
mg/L
  Day 1, pre-breakfast: number analyzed (Participants) | 4 | 3 | 3 | 3 | 5
  Day 1, pre-breakfast | 15.3 (11.30) | 17.7 (11.50) | 8.7 (5.51) | 15.7 (8.33) | 6.6 (0.89)
  Day 7, pre-breakfast: number analyzed (Participants) | 3 | 4 | 2 | 6 | 3
  Day 7, pre-breakfast | 8.0 (1.73) | 19.5 (27.67) | 24.5 (20.51) | 24.0 (22.60) | 7.3 (1.53)
  Day 14, 24 hours: number analyzed (Participants) | 4 | 3 | 5 | 4 | 5
  Day 14, 24 hours | 7.8 (2.50) | 28.3 (34.53) | 11.4 (6.31) | 11.0 (3.56) | 10.4 (8.88)
  Follow up: number analyzed (Participants) | 6 | 8 | 9 | 2 | 5
  Follow up | 54.0 (78.01) | 26.1 (35.34) | 17.6 (13.87) | 29.5 (34.65) | 11.2 (5.17)

11. Primary Outcome: Mean Value of Urine pH (Part A)
Description: Urine samples were collected at screening, Day -1, at 24hr post- dose (Day 2), and at follow-up. Urinalysis parameters included urine pH assessed using dipstick analysis. pH is calculated on a scale of 0 to 14, such that, the lower the number, more acidic the urine and higher the number, more alkaline the urine with 7 being neutral.
Time Frame: Up to 10 days after discharge (Day 2) in Part A
Population: Safety Population
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part A
Number analyzed (Participants) | 6
pH
  Day 1, 24 hours | 6.17 (0.258)
  Follow up | 5.92 (0.376)

12. Primary Outcome: Mean Value of Urine pH (Part B)
Description: Urine samples were collected at screening, on Day -2, and on Days 1, 7, 15 and at follow-up. Urinalysis parameters included urine pH assessed using dipstick analysis. pH is calculated on a scale of 0 to 14, such that, the lower the number, more acidic the urine and higher the number, more alkaline the urine with 7 being neutral.
Time Frame: Up to 10 days after discharge (Day 15) in Part B
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 15 | 13
pH
  Day 1, pre-breakfast | 6.04 (0.499) | 6.04 (0.431) | 6.04 (0.257) | 6.03 (0.399) | 5.92 (0.344)
  Day 7, pre-breakfast | 6.11 (0.446) | 5.85 (0.240) | 6.00 (0.369) | 6.07 (0.458) | 6.04 (0.380)
  Day 14, 24 hours: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 14, 24 hours | 5.96 (0.414) | 6.04 (0.247) | 6.17 (0.326) | 6.07 (0.267) | 6.08 (0.277)
  Follow up: number analyzed (Participants) | 13 | 12 | 12 | 13 | 12
  Follow up | 6.15 (0.747) | 5.88 (0.483) | 5.96 (0.396) | 6.08 (0.572) | 5.88 (0.311)

13. Primary Outcome: Mean Value of Urine Specific Gravity (Part A)
Description: Urine samples were collected at screening, Day -1, at 24hr post- dose (Day 2), and at follow-up. Urinalysis parameter include urine specific gravity. Urinary specific gravity is a measure of the concentration of solutes in the urine . It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine .
Time Frame: Up to 10 days after discharge (Day 2) in Part A
Population: Safety Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Arm A
Number analyzed (Participants) | 5
Ratio
  Day 1, 24 hours | 1.0150 (0.00500)
  Follow up | 1.0210 (0.00224)

14. Primary Outcome: Mean Value of Urine Specific Gravity (Part B)
Description: Urine samples were collected at screening, on Day -2, and on Days 1, 7, 15 and at follow-up. Urinalysis parameter include urine specific gravity. Urinary specific gravity is a measure of the concentration of solutes in the urine . It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine .
Time Frame: Up to 10 days after discharge (Day 15) in Part B
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 15 | 13
Ratio
  Day 1, pre-breakfast: number analyzed (Participants) | 11 | 8 | 6 | 11 | 10
  Day 1, pre-breakfast | 1.0127 (0.00518) | 1.0144 (0.00417) | 1.0125 (0.00418) | 1.0132 (0.00513) | 1.0135 (0.00580)
  Day 7, pre-breakfast: number analyzed (Participants) | 9 | 11 | 6 | 14 | 11
  Day 7, pre-breakfast | 1.0144 (0.00464) | 1.0177 (0.00564) | 1.0150 (0.00447) | 1.0125 (0.00380) | 1.0141 (0.00539)
  Day 14, 24 hours: number analyzed (Participants) | 10 | 9 | 7 | 11 | 12
  Day 14, 24 hours | 1.0170 (0.00587) | 1.0161 (0.00651) | 1.0143 (0.00607) | 1.0127 (0.00410) | 1.0138 (0.00433)
  Follow up: number analyzed (Participants) | 9 | 8 | 10 | 9 | 10
  Follow up | 1.0200 (0.00661) | 1.0163 (0.00443) | 1.0185 (0.00669) | 1.0172 (0.00618) | 1.0165 (0.00669)

15. Primary Outcome: Number of Participants With Abnormal Vital Signs of PCI (Part A)
Description: Assessment of vital signs (including systolic, diastolic blood pressure and heart rate) was performed at one time point at Screening, at follow-up and pre-breakfast on Day -1. On Day 1, they were taken at pre-breakfast, 1 hour, 3, 4, 6, 10, 16 and 24 hours post-dose. Assessments were made in triplicate at the pre-breakfast time point, and single assessments were made at all other times. Assessments were performed after resting in a supine or semi-supine position for at least 10 minutes. PCI value of systolic blood pressure: <85 and >160 millimeter of mercury (mmHg). PCI value of diastolic blood pressure: <45 and >100 mmHg. PCI value of heart rate: <40 and >110 beats per minute.
Time Frame: Up to 10 days after discharge (Day 2) in Part A
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 6
Participants
  Blood pressure (systolic and diastolic) | 0
  Heart rate, high | 1

16. Primary Outcome: Number of Participants With Abnormal Vital Signs of PCI (Part B)
Description: Assessment of vital signs (including systolic and diastolic blood pressure and heart rate) was performed at Screening, pre-breakfast on Days -1 to 14 in a fasting state early in the morning (prior to morning dosing on Days 1-14), and at Follow-up. On Days 1, 7 and 14, they were taken at 1, 3, 6, 9, 12 and 24 hours after the morning dose. At each time point, assessment was performed after resting in a supine or semi-supine position for at least 10 minutes.
Time Frame: Up to 10 days after discharge (Day 15) in Part B
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 15 | 13
Participants
  Systolic blood pressure, high | 0 | 0 | 1 | 0 | 0
  Heart rate | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings (Part A)
Description: ECGs were taken at Screening, pre-breakfast on Day -1, on Day 1 (pre-breakfast, 1 hour, 2, 3, 4, 6, 8, 13, 24hours post-dose), and at follow-up. Assessments were made in triplicate on Day 1 at the pre-breakfast time point, and single assessments were made at all other times. ECGs were taken in supine position. The data has been presented as abnormal- not clinically significant (NCS) and abnormal-clinically significant (CS).
Time Frame: Up to 10 days after discharge (Day 2) in Part A
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A
Number analyzed (Participants) | 6
Participants
  Day 1, pre-breakfast 1, abnormal-NCS | 3
  Day 1, pre-breakfast 2, abnormal-NCS | 2
  Day 1, pre-breakfast 3, abnormal-NCS | 2
  Day 1, 1 hour, abnormal-NCS | 1
  Day 1, 2 hour, abnormal-NCS | 3
  Day 1, 3 hour, abnormal-NCS | 3
  Day 1, 4 hour, abnormal-NCS | 2
  Day 1, 6 hour, abnormal-NCS | 1
  Day 1, 8 hour, abnormal-NCS | 3
  Day 1, 13 hour, abnormal-NCS | 1
  Day 1, 24 hour, abnormal-NCS | 2

18. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings (Part B)
Description: ECGs were taken at Screening, pre-breakfast on Day -1 and at Follow-up. On Days 1, 7 and 14 ECGs were taken pre-breakfast (fasting) and at 1, 2, 4, 6, 8, 12 and 24hours post-dose. Triplicate ECGs were taken at the pre-breakfast time point, and single assessments were taken at all other times. ECGs were taken in supine position. The data has been presented as abnormal- not clinically significant (NCS) and abnormal-clinically significant (CS).
Time Frame: Up to 10 days after discharge (Day 15) in Part B
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 15 | 13
Participants
  Day 1, pre-breakfast 1, abnormal-NCS | 2 | 2 | 4 | 3 | 3
  Day 1, pre-breakfast 2, abnormal-NCS | 1 | 2 | 5 | 2 | 4
  Day 1, pre-breakfast 3, abnormal-NCS | 1 | 2 | 5 | 2 | 4
  Day 1, 1 hour, abnormal-NCS | 1 | 1 | 4 | 6 | 3
  Day 1, 1 hour, abnormal-CS | 0 | 1 | 0 | 0 | 0
  Day 1, 2 hour, abnormal-NCS | 1 | 1 | 3 | 4 | 2
  Day 1, 4 hour, abnormal-NCS | 1 | 2 | 4 | 4 | 2
  Day 1, 6 hour, abnormal-NCS | 2 | 2 | 4 | 4 | 3
  Day 1, 8 hour, abnormal-NCS | 1 | 4 | 4 | 4 | 3
  Day 1, 12 hour, abnormal-NCS | 1 | 3 | 3 | 3 | 3
  Day 1, 24 hour, abnormal-NCS | 3 | 2 | 3 | 3 | 4
  Day 7, pre-breakfast 1, abnormal-NCS | 1 | 2 | 4 | 3 | 3
  Day 7, pre-breakfast 2, abnormal-NCS | 2 | 3 | 4 | 3 | 2
  Day 7, pre-breakfast 3, abnormal-NCS | 1 | 3 | 3 | 2 | 3
  Day 7, 1 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 7, 1 hour, abnormal-NCS | 0 | 1 | 5 | 2 | 4
  Day 7, 2 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 7, 2 hour, abnormal-NCS | 0 | 3 | 5 | 3 | 3
  Day 7, 4 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 7, 4 hour, abnormal-NCS | 0 | 2 | 4 | 3 | 4
  Day 7, 6 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 7, 6 hour, abnormal-NCS | 0 | 3 | 3 | 2 | 5
  Day 7, 8 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 7, 8 hour, abnormal-NCS | 1 | 4 | 4 | 2 | 3
  Day 7, 12 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 7, 12 hour, abnormal-NCS | 2 | 2 | 3 | 2 | 3
  Day 7, 24 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 7, 24 hour, abnormal-NCS | 1 | 3 | 4 | 3 | 4
  Day 14, pre-breakfast 1, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 14, pre-breakfast 1, abnormal-NCS | 1 | 1 | 4 | 3 | 4
  Day 14, pre-breakfast 2, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 14, pre-breakfast 2, abnormal-NCS | 1 | 2 | 5 | 3 | 4
  Day 14, pre-breakfast 3, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 14, pre-breakfast 3, abnormal-NCS | 1 | 1 | 4 | 3 | 4
  Day 14, 1 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 14, 1 hour, abnormal-NCS | 1 | 3 | 5 | 2 | 2
  Day 14, 2 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 14, 2 hour, abnormal-NCS | 1 | 2 | 4 | 3 | 2
  Day 14, 4 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 14, 4 hour, abnormal-NCS | 0 | 2 | 3 | 3 | 3
  Day 14, 6 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 14, 6 hour, abnormal-NCS | 0 | 2 | 4 | 2 | 1
  Day 14, 8 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 12
  Day 14, 8 hour, abnormal-NCS | 1 | 1 | 0 | 1 | 1
  Day 14, 12 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 12
  Day 14, 12 hour, abnormal-NCS | 1 | 2 | 5 | 3 | 2
  Day 14, 24 hour, abnormal-NCS: number analyzed (Participants) | 14 | 13 | 12 | 14 | 13
  Day 14, 24 hour, abnormal-NCS | 1 | 1 | 5 | 3 | 3
  Follow up-NCS | 1 | 2 | 2 | 3 | 3

19. Primary Outcome: Area Under the Concentration-time Curve From Zero (Pre-dose) to 24 Hours [AUC (0-24)] and AUC From Time Zero (Pre-dose) to Last Time of Quantifiable Concentration (AUC [0-last)] Following a Single Dose of GSK1292263 (Part A)
Description: Blood samples for the determination of pharmacokinetics (PK) were collected on Day 1 Immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13, 24 and 48 hours post-dose. PK samples for 2 participants were not analyzed. The PK parameters were calculated by standard non-compartmental analysis. AUC (0-last) and AUC (0-24) were determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: On Day 1 Immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13, 24 and 48 hours post-dose.
Population: The PK Population included participants from the Safety Population who had any PK parameter estimated. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms hour per milliliter (ng*hr/mL)
Arm/Group | Part A
Number analyzed (Participants) | 4
nanograms hour per milliliter (ng*hr/mL)
  AUC (0-24) | 7046.25 (11.090)
  AUC (0-last) | 10099.35 (14.332)

20. Primary Outcome: Maximum Observed Concentration (Cmax) Following a Single Dose of GSK1292263 (Part A)
Description: Blood samples for the determination of PK were collected on Day 1 Immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13, 24 and 48 hours post-dose. PK samples for participants were not analyzed. The PK parameters were calculated by standard non-compartmental analysis. Cmax was determined directly from the raw concentration-time data.
Time Frame: On Day 1 Immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13, 24 and 48 hours post-dose.
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part A
Number analyzed (Participants) | 4
nanograms per milliliter (ng/mL) | 582.619 (28.0710)

21. Primary Outcome: Lag Time Before Observation of Drug Concentrations in Sampled Matrix (Tlag) and Time of Occurrence of Cmax (Tmax) Following a Single Dose of GSK1292263 (Part A)
Description: Blood samples for the determination of PK were collected on Day 1 Immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13, 24 and 48 hours post-dose. PK samples for 2 participants were not analyzed. The PK parameters were calculated by standard non-compartmental analysis. Tmax was determined directly from the raw concentration-time data. Tlag was determined as the time of the sample preceding the first quantifiable concentration, on Day 1 only.
Time Frame: On Day 1 Immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13, 24 and 48 hours post-dose.
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: hour
Arm/Group | Part A
Number analyzed (Participants) | 4
hour
  Tlag | 0.000 [0.00 to 0.50]
  Tmax | 5.00 [4.0 to 13.0]

22. Primary Outcome: Apparent Clearance Following Oral Dosing (CL/F) of GSK1292263 (Part A)
Description: Outcome measure was added with caveat "as data permits". The data for CL/F was not collected.
Time Frame: On Day 1 Immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13, 24 and 48 hours post-dose.
Arm/Group | Part A
Number analyzed (Participants) | 0

23. Primary Outcome: Volume of Distribution (V/F) (Part A)
Description: Outcome measure was added with caveat "as data permits". The data for V/F was not collected.
Time Frame: On Day 1 Immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13, 24 and 48 hours post-dose.
Population: PK Population
Arm/Group | Part A
Number analyzed (Participants) | 0

24. Primary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC [0-inf]) Following a Single Dose of GSK1292263 (Part A)
Description: Outcome measure was added with caveat "as data permits". The data for AUC (0-inf) was not collected.
Time Frame: On Day 1 Immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13, 24 and 48 hours post-dose.
Population: PK Population
Arm/Group | Part A
Number analyzed (Participants) | 0

25. Primary Outcome: Terminal Phase Half-life (t1/2) Following a Single Dose of GSK1292263 (Part A)
Description: Outcome measure was added with caveat "as data permits". The data for t1/2 was not collected.
Time Frame: On Day 1 Immediately pre-dose (time 0) and at 0.5, 1, 2, 3, 4, 6, 8, 13, 24 and 48 hours post-dose.
Population: PK Population
Arm/Group | Part A
Number analyzed (Participants) | 0

26. Primary Outcome: Cmax Following Repeat Dose of GSK1292263 (Part B)
Description: Serial blood samples for the determination of the PK of GSK1292263 were collected on Days 1, 7 and 14. Blood samples for PK were collected on Days 1 and 14, at immediately pre-morning dose, 1, 2, 4, 6, 8, 10, 11, 12, 14, 16, 18, 24 and 48 hours post-morning dose. On Day 7, blood samples for PK were collected at pre-dose (post-breakfast), 1, 2, 4 (pre-lunch), 6 and 10 (immediately post-dinner, pre-dose for BID regimen). When planned PK sampling resulted in multiple samples at the same time point, only one sample was collected. The PK parameters were calculated by standard non-compartmental analysis. Cmax was determined directly from the raw concentration-time data.
Time Frame: On Days 1 and 14, at immediately pre-morning dose, 1, 2, 4, 6, 8, 10, 11, 12, 14, 16, 18, 24 and 48 hours post-morning dose. On Day 7, at pre-dose (post-breakfast), 1, 2, 4 (pre-lunch), 6 and 10 (immediately post-dinner, pre-dose for BID regimen).
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg
Number analyzed (Participants) | 13 | 12 | 15
ng/mL
  Day 1 | 278.451 (36.5951) | 686.845 (33.1747) | 610.586 (29.2427)
  Day 7: number analyzed (Participants) | 13 | 12 | 14
  Day 7 | 416.441 (30.0099) | 872.843 (22.2509) | 738.918 (39.1209)
  Day 14: number analyzed (Participants) | 13 | 12 | 14
  Day 14 | 457.716 (20.4386) | 902.325 (30.0011) | 664.505 (37.8497)

27. Primary Outcome: Tmax and Tlag Following Repeat Dose of GSK1292263 (Part B)
Description: Serial blood samples for the determination of the PK of GSK1292263 were collected on Days 1, 7 and 14. Blood samples for PK were collected on Days 1 and 14, at immediately pre-morning dose, 1, 2, 4, 6, 8, 10, 11, 12, 14, 16, 18, 24 and 48 hours post-morning dose. On Day 7, blood samples for PK were collected at pre-dose (post-breakfast), 1, 2, 4 (pre-lunch), 6 and 10 (immediately post-dinner, pre-dose for BID regimen). When planned PK sampling resulted in multiple samples at the same time point, only one sample was collected. The PK parameters were calculated by standard non-compartmental analysis. Tmax was determined directly from the raw concentration-time data. Tlag was determined as the time of the sample preceding the first quantifiable concentration, on Day 1 only.
Time Frame: as for outcome 26
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Median (Full Range); unit: hour
Arm/Group | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg
Number analyzed (Participants) | 13 | 12 | 15
hour
  Tlag, Day1 | 0.000 [0.00 to 1.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 1.00]
  Tmax, Day 1 | 14.00 [6.0 to 18.0] | 14.00 [4.0 to 18.0] | 4.0 [4.0 to 12.0]
  Tmax, Day 7: number analyzed (Participants) | 13 | 12 | 14
  Tmax, Day 7 | 4.00 [4.0 to 6.0] | 4.00 [0.0 to 4.0] | 4.00 [2.0 to 10.1]
  Tmax, Day 14 | 4.00 [4.0 to 24.0] | 13.00 [1.0 to 24.0] | 4.0 [1.0 to 10.2]

28. Primary Outcome: AUC From Time Zero (Pre-dose) to 10 Hours [AUC (0-10)] and AUC (0-24) Following Repeat Dose of GSK1292263 (Part B)
Description: Serial blood samples for the determination of the PK of GSK1292263 were collected on Days 1, 7 and 14. Blood samples for PK were collected on Days 1 and 14, at immediately pre-morning dose, 1, 2, 4, 6, 8, 10, 11, 12, 14, 16, 18, 24 and 48 hours post-morning dose. On Day 7, blood samples for PK were collected at pre-dose (post-breakfast), 1, 2, 4 (pre-lunch), 6 and 10 (immediately post-dinner, pre-dose for BID regimen). When planned PK sampling resulted in multiple samples at the same time point, only one sample was collected. The PK parameters were calculated by standard non-compartmental analysis. AUC (0-10) and AUC (0-24) were determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: as for outcome 26
Population: PK Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg
Number analyzed (Participants) | 13 | 12 | 15
ng*hr/mL
  AUC (0-10), Day 1 | 1143.35 (36.439) | 3149.94 (38.937) | NA (NA) — Data was not analyzed at this time point
  AUC (0-10), Day 7: number analyzed (Participants) | 13 | 12 | 14
  AUC (0-10), Day 7 | 2930.47 (21.366) | 6472.68 (29.790) | 5205.86 (31.529)
  AUC (0-10), Day 14 | 3130.50 (22.430) | 6057.41 (32.784) | NA (NA) — Data was not analyzed at this time point
  AUC (0-24), Day 1 | 3775.76 (30.915) | 9968.88 (39.959) | 6791.90 (24.550)
  AUC (0-24), Day 14: number analyzed (Participants) | 13 | 12 | 14
  AUC (0-24), Day 14 | 7785.24 (19.152) | 15479.48 (33.009) | 9391.30 (32.948)

29. Primary Outcome: T1/2 Following Repeat Dose of GSK1292263 (Part B)
Description: Outcome measure was added with caveat "as data permits". The data for T1/2 was not collected.
Time Frame: as for outcome 26
Population: PK population
Arm/Group | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg
Number analyzed (Participants) | 0 | 0 | 0

30. Primary Outcome: Mean Accumulation Ratio by AUC (0-10), AUC (0-24) and Cmax for GSK1292263 (Part B)
Description: Accumulation ratio (Ro) was derived as: Ro = Day 14 morning AUC(0-10)/Day 1 morning AUC(0-10) (for BID regimens only). Ro = Day 14 AUC(0-24)/Day 1 AUC(0-24) (for both BID and once daily regimens). Accumulation ratio (RCmax)= Day 14 Cmax/Day 1 Cmax. RCmax was not computed for each dosing period (morning and evening).
Time Frame: On Days 1 and 14, at immediately pre-morning dose, 1, 2, 4, 6, 8, 10, 11, 12, 14, 16, 18, 24 and 48 hours post-morning dose.
Population: PK Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (90% Confidence Interval); unit: Ratio
Arm/Group | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg
Number analyzed (Participants) | 13 | 12 | 14
Ratio
  AUC (0-10) | 2.7380 [2.4706 to 3.0344] | 1.9230 [1.6883 to 2.1903] | NA [NA to NA] — Data was not analyzed at this time point
  AUC (0-24) | 2.0619 [1.8432 to 2.3065] | 1.5528 [1.3748 to 1.7538] | 1.3730 [1.2219 to 1.5429]
  Cmax | 1.6438 [1.4256 to 1.8954] | 1.3137 [1.2009 to 1.4372] | 1.1077 [0.9659 to 1.2704]

31. Primary Outcome: Change From Baseline in Mean Fasted Glucose Value (Part A)
Description: Baseline was considered to be Day 1 pre-breakfast. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline is set to missing as well. If measurements were taken in triplicate, then the mean of the triplicate measurements was used as the Baseline.
Time Frame: Baseline and at pre-breakfast on Day 1 and 24 h post-dose.
Population: The Pharmacodynamic (PD) Population included participants from the Safety Population who had any PD parameter estimated. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millimoles per liter (mmol/L)
Arm/Group | Part A
Number analyzed (Participants) | 4
millimoles per liter (mmol/L) | 0.17 (-199.736)

32. Primary Outcome: Change From Baseline in Mean Fasted Insulin Value (Part A)
Description: as for outcome 31
Time Frame: Baseline and at pre-breakfast on Day 1 and 24 hours post-dose.
Population: PD Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles per liter (pmol/L)
Arm/Group | Part A
Number analyzed (Participants) | 4
picomoles per liter (pmol/L) | 3.45 (-187.128)

33. Primary Outcome: Change From Baseline in Mean Fasted Glucose Value (Part B)
Description: Baseline was considered to be Day -1 pre-breakfast value. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline is set to missing as well. If measurements were taken in triplicate, then the mean of the triplicate measurements was used as the Baseline.
Time Frame: Baseline and at pre-breakfast on Days -1 and 14, and then at 0.5, 1, 1.5, 2 and 3 hours post dose.
Population: PD Population.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 14 | 12
mmol/L
  Day 7, pre-breakfast | -0.53 [-0.92 to -0.14] | -0.74 [-1.22 to -0.27] | -0.28 [-1.15 to 0.58] | 0.21 [-0.53 to 0.95] | -1.75 [-2.20 to -1.29]
  Day 14, pre-breakfast | -0.74 [-1.30 to -0.18] | -1.57 [-2.39 to -0.75] | -0.81 [-1.77 to 0.16] | -0.11 [-0.96 to 0.75] | -1.83 [-2.65 to -1.02]
  Day 14, 24 hours | -0.01 [-0.94 to 0.92] | -0.57 [-1.49 to 0.36] | 0.66 [-0.31 to 1.64] | 0.68 [0.09 to 1.27] | -1.06 [-1.87 to -0.26]
Statistical Analysis 1: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -0.216, 95% CI 2-sided [-1.00 to 0.57]
Statistical Analysis 2: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 0.290, 95% CI 2-sided [-0.53 to 1.11]
Statistical Analysis 3: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 0.748, 95% CI 2-sided [-0.02 to 1.52]
Statistical Analysis 4: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -1.207, 95% CI 2-sided [-2.01 to -0.41]
Statistical Analysis 5: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Day 7 , pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 0.991, 95% CI 2-sided [0.18 to 1.81]
Statistical Analysis 6: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 1.497, 95% CI 2-sided [0.66 to 2.34]
Statistical Analysis 7: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 1.955, 95% CI 2-sided [1.16 to 2.75]
Statistical Analysis 8: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -0.780, 95% CI 2-sided [-1.74 to 0.18]
Statistical Analysis 9: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 0.188, 95% CI 2-sided [-0.81 to 1.19]
Statistical Analysis 10: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 0.600, 95% CI 2-sided [-0.35 to 1.55]
Statistical Analysis 11: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -1.069, 95% CI 2-sided [-2.05 to -0.08]
Statistical Analysis 12: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 0.289, 95% CI 2-sided [-0.71 to 1.29]
Statistical Analysis 13: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 1.257, 95% CI 2-sided [0.22 to 2.29]
Statistical Analysis 14: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 1.669, 95% CI 2-sided [0.68 to 2.65]
Statistical Analysis 15: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = -0.556, 95% CI 2-sided [-1.65 to 0.54]
Statistical Analysis 16: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = 0.745, 95% CI 2-sided [-0.40 to 1.89]
Statistical Analysis 17: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = 0.711, 95% CI 2-sided [-0.36 to 1.78]
Statistical Analysis 18: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = -1.030, 95% CI 2-sided [-2.15 to 0.09]
Statistical Analysis 19: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = 0.474, 95% CI 2-sided [-0.66 to 1.61]
Statistical Analysis 20: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = 1.775, 95% CI 2-sided [0.60 to 2.95]
Statistical Analysis 21: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = 1.741, 95% CI 2-sided [0.63 to 2.86]

34. Primary Outcome: Change From Baseline in Mean Fasted Insulin Value (Part B)
Description: as for outcome 33
Time Frame: Baseline and at pre-breakfast on Days -1 and 14, and then at 0.5, 1, 1.5, 2 and 3 hours post dose.
Population: PD Population.
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 14 | 12
pmol/L
  Day 7, pre-breakfast | -2.74 [-15.26 to 9.77] | -1.84 [-9.22 to 5.53] | -26.34 [-57.25 to 4.57] | -22.99 [-39.68 to -6.31] | 2.07 [-15.96 to 20.11]
  Day 14, pre-breakfast | 4.84 [-8.97 to 18.65] | 6.22 [-5.01 to 17.46] | -13.48 [-36.79 to 9.82] | -33.26 [-53.15 to -13.37] | 4.43 [-5.65 to 14.50]
  Day 14, 24 hours | 23.25 [5.53 to 40.96] | 4.97 [-19.94 to 29.87] | -12.54 [-40.87 to 15.80] | -17.52 [-41.26 to 6.23] | 27.47 [2.50 to 52.43]
Statistical Analysis 1: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 0.195, 95% CI 2-sided [-17.17 to 17.56]
Statistical Analysis 2: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -16.863, 95% CI 2-sided [-34.70 to 0.98]
Statistical Analysis 3: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -5.460, 95% CI 2-sided [-23.04 to 12.12]
Statistical Analysis 4: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 3.850, 95% CI 2-sided [-13.89 to 21.58]
Statistical Analysis 5: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -3.655, 95% CI 2-sided [-21.70 to 14.39]
Statistical Analysis 6: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -20.712, 95% CI 2-sided [-39.25 to -2.17]
Statistical Analysis 7: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Day 7, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -9.310, 95% CI 2-sided [-27.63 to 9.01]
Statistical Analysis 8: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -3.649, 95% CI 2-sided [-19.43 to 12.14]
Statistical Analysis 9: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -16.660, 95% CI 2-sided [-32.72 to -0.60]
Statistical Analysis 10: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -22.251, 95% CI 2-sided [-38.34 to -6.16]
Statistical Analysis 11: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -4.590, 95% CI 2-sided [-20.69 to 11.51]
Statistical Analysis 12: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = 0.941, 95% CI 2-sided [-15.40 to 17.28]
Statistical Analysis 13: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -12.070, 95% CI 2-sided [-28.82 to 4.68]
Statistical Analysis 14: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Day 14, pre-breakfast; Test type: Superiority or Other; Mean Difference (Net) = -17.662, 95% CI 2-sided [-34.72 to -0.60]
Statistical Analysis 15: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = -19.101, 95% CI 2-sided [-44.00 to 5.80]
Statistical Analysis 16: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = -27.976, 95% CI 2-sided [-53.56 to -2.39]
Statistical Analysis 17: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = -23.609, 95% CI 2-sided [-48.82 to 1.60]
Statistical Analysis 18: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = 3.094, 95% CI 2-sided [-22.34 to 28.53]
Statistical Analysis 19: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = -22.194, 95% CI 2-sided [-48.07 to 3.69]
Statistical Analysis 20: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = -31.070, 95% CI 2-sided [-57.66 to -4.48]
Statistical Analysis 21: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Day 14, 24 hours; Test type: Superiority or Other; Mean Difference (Net) = -26.703, 95% CI 2-sided [-52.98 to -0.42]

35. Primary Outcome: Mean Post Meal Glucose Value (Part B)
Description: Blood samples were collected on Days -1 and 14, post-breakfast at 0.5, 1, 1.5, 2 and 3 hours post dose. For lunch (approximately 4 hours post morning dose) samples were collected at the following times after starting each meal: 0.5, 1, 1.5, 2 and 3 hours. For the evening meal (approximately 10 hours post morning dose), samples were taken at 0.5, 1, 1.5, 2 and 3 hours post dinner.
Time Frame: At pre-breakfast on Days -1 and 14, and then at 0.5, 1, 1.5, 2 and 3 hours post dose.
Population: PD Population.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 14 | 12
mmol/L
  Day -1, post-breakfast, 0.5 hour | 13.75 [12.80 to 14.70] | 13.51 [12.35 to 14.67] | 14.68 [13.74 to 15.62] | 13.04 [11.67 to 14.42] | 13.60 [12.63 to 14.56]
  Day -1, post-breakfast, 1 hour | 13.62 [12.58 to 14.66] | 13.42 [12.39 to 14.45] | 14.48 [13.49 to 15.48] | 13.43 [12.06 to 14.80] | 13.12 [11.88 to 14.37]
  Day -1, post-breakfast, 1.5 hour | 12.56 [11.41 to 13.71] | 12.12 [10.90 to 13.34] | 12.94 [11.62 to 14.26] | 12.02 [10.24 to 13.80] | 11.39 [10.17 to 12.60]
  Day -1, post-breakfast, 2 hour | 10.71 [9.73 to 11.69] | 10.55 [9.03 to 12.06] | 11.50 [9.99 to 13.01] | 10.67 [9.04 to 12.29] | 9.75 [8.46 to 11.03]
  Day -1, post-breakfast, 3 hour | 7.78 [7.02 to 8.53] | 8.48 [6.68 to 10.28] | 8.68 [7.02 to 10.33] | 8.46 [6.99 to 9.93] | 7.73 [6.91 to 8.55]
  Day -1, post-lunch, 0.5 hour | 7.46 [6.48 to 8.45] | 8.90 [7.35 to 10.45] | 8.56 [7.54 to 9.58] | 8.58 [7.61 to 9.56] | 7.93 [7.04 to 8.83]
  Day -1, post-lunch, 1 hour | 10.31 [9.47 to 11.15] | 11.19 [10.09 to 12.29] | 10.71 [9.85 to 11.57] | 10.12 [8.76 to 11.48] | 10.36 [9.34 to 11.39]
  Day -1, post-lunch, 1.5 hour | 11.07 [9.99 to 12.14] | 11.17 [9.75 to 12.58] | 11.64 [10.54 to 12.74] | 10.45 [9.02 to 11.89] | 10.69 [9.51 to 11.87]
  Day -1, post-lunch, 2 hour | 11.31 [10.11 to 12.51] | 10.82 [9.42 to 12.21] | 11.75 [10.72 to 12.78] | 10.11 [8.82 to 11.39] | 10.72 [9.56 to 11.88]
  Day -1, post-lunch, 3 hour | 11.05 [9.95 to 12.16] | 10.05 [8.50 to 11.60] | 11.25 [10.08 to 12.43] | 10.37 [9.03 to 11.71] | 9.92 [8.80 to 11.03]
  Day -1, post-dinner, 0.5 hour | 9.28 [7.95 to 10.60] | 9.19 [8.14 to 10.25] | 8.78 [7.85 to 9.71] | 8.92 [7.86 to 9.98] | 8.39 [7.56 to 9.22]
  Day -1, post-dinner, 1 hour | 11.15 [9.83 to 12.47] | 11.27 [9.88 to 12.67] | 11.00 [9.75 to 12.25] | 10.77 [9.64 to 11.90] | 10.27 [9.33 to 11.22]
  Day -1, post-dinner, 1.5 hour | 11.45 [10.13 to 12.77] | 10.97 [9.46 to 12.49] | 10.99 [9.97 to 12.01] | 10.94 [9.62 to 12.26] | 10.52 [9.47 to 11.58]
  Day -1, post-dinner, 2 hour | 11.67 [10.15 to 13.20] | 10.76 [9.18 to 12.35] | 10.81 [9.76 to 11.85] | 10.98 [9.57 to 12.39] | 10.18 [9.09 to 11.27]
  Day -1, post-dinner, 3 hour | 11.58 [9.76 to 13.39] | 10.41 [8.83 to 11.99] | 10.34 [9.45 to 11.23] | 10.48 [9.20 to 11.75] | 9.66 [8.49 to 10.84]
  Day 14, post-breakfast, 0.5 hour | 14.16 [12.45 to 15.86] | 13.13 [11.86 to 14.41] | 14.96 [13.89 to 16.03] | 13.83 [12.60 to 15.05] | 12.26 [10.53 to 13.98]
  Day 14, post-breakfast, 1 hour | 14.02 [11.79 to 16.24] | 13.32 [11.47 to 15.17] | 14.23 [12.91 to 15.55] | 14.32 [12.95 to 15.70] | 12.03 [10.17 to 13.89]
  Day 14, post-breakfast, 1.5 hour | 12.69 [11.25 to 14.13] | 11.58 [9.63 to 13.52] | 12.96 [11.14 to 14.78] | 13.07 [11.37 to 14.76] | 10.55 [8.66 to 12.43]
  Day 14, post-breakfast, 2 hour | 11.15 [9.83 to 12.46] | 9.98 [8.03 to 11.93] | 10.93 [9.10 to 12.76] | 11.11 [9.20 to 13.02] | 9.10 [7.21 to 11.00]
  Day 14, post-breakfast, 3 hour | 7.56 [6.14 to 8.98] | 6.96 [5.32 to 8.61] | 8.20 [6.58 to 9.82] | 8.73 [7.04 to 10.43] | 6.69 [5.06 to 8.32]
  Day 14, post-lunch, 0.5 hour | 7.43 [6.43 to 8.44] | 8.73 [7.66 to 9.80] | 10.07 [8.84 to 11.31] | 8.70 [7.76 to 9.63] | 7.77 [6.66 to 8.89]
  Day 14, post-lunch, 1 hour | 9.61 [8.42 to 10.80] | 10.59 [9.29 to 11.88] | 11.96 [10.62 to 13.29] | 10.42 [9.24 to 11.59] | 8.38 [7.47 to 9.28]
  Day 14, post-lunch, 1.5 hour | 10.38 [9.23 to 11.53] | 10.80 [9.43 to 12.17] | 12.33 [11.25 to 13.41] | 11.12 [9.69 to 12.55] | 8.83 [7.78 to 9.88]
  Day 14, post-lunch, 2 hour | 10.83 [9.25 to 12.40] | 10.51 [9.15 to 11.88] | 12.09 [10.85 to 13.33] | 10.87 [9.48 to 12.27] | 8.84 [7.78 to 9.91]
  Day 14, post-lunch, 3 hour | 10.51 [8.71 to 12.30] | 9.71 [8.03 to 11.40] | 10.57 [9.12 to 12.01] | 10.44 [8.91 to 11.96] | 8.90 [7.76 to 10.05]
  Day 14, post-dinner, 0.5 hour | 8.17 [6.86 to 9.47] | 7.99 [6.95 to 9.03] | 9.37 [8.09 to 10.65] | 10.41 [8.96 to 11.86] | 7.29 [6.40 to 8.19]
  Day 14, post-dinner, 1 hour | 11.07 [9.53 to 12.61] | 11.20 [10.03 to 12.36] | 12.21 [10.72 to 13.70] | 12.56 [10.99 to 14.12] | 9.43 [8.00 to 10.86]
  Day 14, post-dinner, 1.5 hour | 11.65 [9.89 to 13.41] | 11.81 [10.43 to 13.19] | 13.01 [11.38 to 14.64] | 13.03 [11.57 to 14.49] | 10.41 [8.48 to 12.33]
  Day 14, post-dinner, 2 hour | 11.42 [9.64 to 13.21] | 11.27 [9.62 to 12.93] | 12.07 [10.76 to 13.38] | 12.60 [11.11 to 14.09] | 10.07 [8.11 to 12.03]
  Day 14, post-dinner, 3 hour | 10.43 [8.77 to 12.10] | 9.78 [7.70 to 11.87] | 10.69 [9.24 to 12.13] | 11.75 [10.17 to 13.32] | 8.80 [7.41 to 10.20]

36. Primary Outcome: Mean Post Meal Insulin Value (Part B)
Description: as for outcome 35
Time Frame: At pre-breakfast on Days -1 and 14, and then at 0.5, 1, 1.5, 2 and 3 hours post dose.
Population: PD Population.
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 14 | 12
pmol/L
  Day -1, post-breakfast, 0.5 hour | 201.81 [120.26 to 283.36] | 185.34 [136.03 to 234.64] | 270.35 [139.59 to 401.11] | 264.15 [183.44 to 344.87] | 219.24 [146.34 to 292.15]
  Day -1, post-breakfast, 1 hour | 222.44 [153.65 to 291.23] | 258.37 [176.77 to 339.98] | 296.05 [161.61 to 430.50] | 338.58 [218.57 to 458.59] | 251.79 [167.51 to 336.07]
  Day -1, post-breakfast, 1.5 hour | 251.01 [161.79 to 340.24] | 246.76 [177.95 to 315.57] | 318.38 [155.32 to 481.44] | 351.10 [239.19 to 463.01] | 237.46 [153.03 to 321.90]
  Day -1, post-breakfast, 2 hour | 233.85 [153.97 to 313.73] | 221.27 [147.26 to 295.28] | 258.69 [108.85 to 408.52] | 304.66 [205.71 to 403.60] | 196.53 [154.15 to 238.91]
  Day -1, post-breakfast, 3 hour | 131.95 [77.37 to 186.53] | 114.67 [85.59 to 143.75] | 162.58 [89.16 to 235.99] | 180.43 [130.54 to 230.32] | 106.98 [69.24 to 144.72]
  Day -1, post-lunch, 0.5 hour | 135.17 [88.11 to 182.22] | 115.21 [68.21 to 162.22] | 147.60 [80.48 to 214.71] | 187.22 [133.25 to 241.19] | 109.63 [85.23 to 134.03]
  Day -1, post-lunch, 1 hour | 193.80 [115.60 to 272.00] | 193.65 [127.73 to 259.57] | 186.02 [113.55 to 258.49] | 246.08 [180.25 to 311.90] | 180.49 [128.88 to 232.10]
  Day -1, post-lunch, 1.5 hour | 188.57 [123.30 to 253.85] | 208.37 [138.94 to 277.80] | 212.29 [135.68 to 288.90] | 289.19 [187.79 to 390.59] | 173.21 [124.34 to 222.08]
  Day -1, post-lunch, 2 hour | 235.41 [106.82 to 363.99] | 196.74 [156.56 to 236.93] | 218.67 [106.48 to 330.87] | 295.21 [185.14 to 405.29] | 202.47 [147.19 to 257.74]
  Day -1, post-lunch, 3 hour | 191.74 [120.96 to 262.51] | 171.15 [120.83 to 221.47] | 207.00 [98.15 to 315.86] | 270.43 [185.95 to 354.91] | 167.37 [125.31 to 209.42]
  Day -1, post-dinner, 0.5 hour | 132.04 [96.91 to 167.16] | 131.50 [81.60 to 181.39] | 150.10 [90.51 to 209.68] | 207.99 [152.25 to 263.72] | 104.16 [77.66 to 130.67]
  Day -1, post-dinner, 1 hour | 199.54 [142.13 to 256.94] | 205.59 [142.87 to 268.31] | 226.22 [127.02 to 325.41] | 274.72 [194.26 to 355.17] | 149.94 [122.06 to 177.81]
  Day -1, post-dinner, 1.5 hour | 195.55 [137.43 to 253.67] | 183.16 [135.87 to 230.46] | 206.80 [119.94 to 293.65] | 275.17 [200.75 to 349.59] | 171.08 [131.77 to 210.38]
  Day -1, post-dinner, 2 hour | 209.64 [130.71 to 288.56] | 205.06 [148.39 to 261.73] | 206.16 [122.43 to 289.88] | 266.34 [184.02 to 348.66] | 171.94 [126.51 to 217.36]
  Day -1, post-dinner, 3 hour | 176.48 [94.31 to 258.66] | 164.28 [110.19 to 218.37] | 172.36 [102.77 to 241.95] | 225.12 [156.84 to 293.39] | 155.62 [110.73 to 200.50]
  Day 14, post-breakfast, 0.5 hour | 258.61 [214.57 to 302.65] | 240.43 [163.71 to 317.15] | 241.13 [163.33 to 318.93] | 259.89 [166.35 to 353.44] | 268.74 [202.79 to 334.70]
  Day 14, post-breakfast, 1 hour | 304.23 [220.12 to 388.34] | 280.93 [201.95 to 359.91] | 297.58 [188.61 to 406.54] | 348.37 [199.81 to 496.92] | 354.57 [253.16 to 455.98]
  Day 14, post-breakfast, 1.5 hour | 297.57 [222.91 to 372.23] | 299.22 [183.56 to 414.89] | 272.63 [201.63 to 343.64] | 409.93 [231.64 to 588.22] | 300.33 [203.08 to 397.57]
  Day 14, post-breakfast, 2 hour | 283.85 [206.65 to 361.06] | 234.65 [167.00 to 302.29] | 229.72 [135.19 to 324.26] | 333.39 [175.19 to 491.60] | 246.53 [176.74 to 316.32]
  Day 14, post-breakfast, 3 hour | 161.67 [91.12 to 232.21] | 110.81 [79.94 to 141.68] | 122.31 [68.67 to 175.94] | 188.31 [120.35 to 256.27] | 117.21 [64.59 to 169.83]
  Day 14, post-lunch, 0.5 hour | 153.65 [104.68 to 202.62] | 129.25 [88.96 to 169.54] | 126.26 [92.54 to 159.98] | 169.17 [122.63 to 215.71] | 155.68 [126.09 to 185.26]
  Day 14, post-lunch, 1 hour | 201.54 [133.12 to 269.95] | 169.74 [130.07 to 209.41] | 172.43 [128.88 to 215.99] | 190.65 [136.34 to 244.96] | 164.53 [133.23 to 195.83]
  Day 14, post-lunch, 1.5 hour | 229.56 [143.82 to 315.30] | 194.93 [141.31 to 248.55] | 179.44 [128.44 to 230.43] | 223.72 [148.81 to 298.63] | 184.69 [145.83 to 223.54]
  Day 14, post-lunch, 2 hour | 237.34 [153.62 to 321.05] | 214.66 [152.23 to 277.09] | 177.88 [131.02 to 224.73] | 227.81 [142.85 to 312.77] | 188.61 [140.47 to 236.75]
  Day 14, post-lunch, 3 hour | 219.31 [111.12 to 327.50] | 181.43 [132.84 to 230.02] | 137.67 [89.10 to 186.24] | 195.64 [140.45 to 250.83] | 172.22 [134.89 to 209.55]
  Day 14, post-dinner, 0.5 hour | 99.41 [60.27 to 138.56] | 98.57 [57.19 to 139.96] | 75.85 [46.65 to 105.04] | 137.16 [100.98 to 173.34] | 92.78 [67.46 to 118.09]
  Day 14, post-dinner, 1 hour | 204.76 [140.32 to 269.19] | 178.38 [129.51 to 227.25] | 141.59 [96.79 to 186.38] | 191.90 [132.03 to 251.77] | 156.48 [119.25 to 193.70]
  Day 14, post-dinner, 1.5 hour | 204.67 [138.63 to 270.71] | 210.90 [150.50 to 271.30] | 163.94 [111.91 to 215.96] | 215.57 [137.16 to 293.98] | 179.94 [140.71 to 219.17]
  Day 14, post-dinner, 2 hour | 237.14 [128.24 to 346.03] | 220.97 [159.61 to 282.32] | 168.71 [100.05 to 237.38] | 223.18 [150.43 to 295.92] | 187.66 [130.14 to 245.19]
  Day 14, post-dinner, 3 hour | 200.85 [106.15 to 295.54] | 167.22 [122.78 to 211.66] | 134.98 [85.91 to 184.05] | 191.01 [133.94 to 248.09] | 175.02 [132.20 to 217.83]

37. Primary Outcome: Change From Baseline in Weighted Mean for Glucose Value (Part B)
Description: Baseline was considered to be Day -1 pre-breakfast value. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline is set to missing as well. If measurements were taken in triplicate, then the mean of the triplicate measurements was used as the Baseline. Weighted mean were assessed for (0-12) and (0-24). AUC with respect to that time interval was calculated using the linear trapezoidal rule. The weighted mean was determined by dividing the AUC by the observed length of the collection interval (time of last assessment - time of first assessment in hours). In order for the AUC to be calculated, the first and last time points and at least one additional assessment falling between the two must be non-missing.
Time Frame: Baseline and at pre-breakfast on Days -1 and 14, and then at 0.5, 1, 1.5, 2 and 3 hours post dose.
Population: PD Population.
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 14 | 12
mmol/L
  Weighted mean (0-12), Day 7 | 0.064 [-0.629 to 0.756] | -0.432 [-1.123 to 0.259] | 0.555 [-0.363 to 1.474] | 1.103 [0.424 to 1.781] | -0.862 [-1.812 to 0.089]
  Weighted mean (0-12), Day 14 | -0.235 [-1.099 to 0.630] | -0.539 [-1.372 to 0.294] | 0.123 [-0.806 to 1.052] | 0.656 [-0.001 to 1.312] | -1.039 [-1.958 to -0.120]
  Weighted mean (0-24), Day 14 | -0.414 [-1.134 to 0.306] | -0.555 [-1.463 to 0.352] | 0.321 [-0.602 to 1.244] | 0.837 [0.126 to 1.548] | -1.025 [-1.889 to -0.161]
Statistical Analysis 1: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = -0.500, 95% CI 2-sided [-1.50 to 0.50]
Statistical Analysis 2: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = 0.513, 95% CI 2-sided [-0.51 to 1.54]
Statistical Analysis 3: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = 1.030, 95% CI 2-sided [0.05 to 2.01]
Statistical Analysis 4: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = -0.955, 95% CI 2-sided [-1.98 to 0.07]
Statistical Analysis 5: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = 0.454, 95% CI 2-sided [-0.59 to 1.50]
Statistical Analysis 6: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = 1.468, 95% CI 2-sided [0.39 to 2.55]
Statistical Analysis 7: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = 1.985, 95% CI 2-sided [0.96 to 3.01]
Statistical Analysis 8: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -0.312, 95% CI 2-sided [-1.38 to 0.76]
Statistical Analysis 9: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = 0.394, 95% CI 2-sided [-0.70 to 1.49]
Statistical Analysis 10: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = 0.875, 95% CI 2-sided [-0.18 to 1.93]
Statistical Analysis 11: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -0.854, 95% CI 2-sided [-1.95 to 0.25]
Statistical Analysis 12: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = 0.542, 95% CI 2-sided [-0.58 to 1.66]
Statistical Analysis 13: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = 1.248, 95% CI 2-sided [0.09 to 2.40]
Statistical Analysis 14: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = 1.729, 95% CI 2-sided [0.63 to 2.83]
Statistical Analysis 15: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -0.148, 95% CI 2-sided [-1.21 to 0.91]
Statistical Analysis 16: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = 0.737, 95% CI 2-sided [-0.34 to 1.81]
Statistical Analysis 17: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = 1.245, 95% CI 2-sided [0.21 to 2.28]
Statistical Analysis 18: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -0.623, 95% CI 2-sided [-1.71 to 0.46]
Statistical Analysis 19: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = 0.475, 95% CI 2-sided [-0.62 to 1.57]
Statistical Analysis 20: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = 1.360, 95% CI 2-sided [0.23 to 2.49]
Statistical Analysis 21: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = 1.869, 95% CI 2-sided [0.79 to 2.95]

38. Primary Outcome: Change From Baseline in Weighted Mean for Insulin Value (Part B)
Description: Baseline was considered to be Day -1 pre-breakfast value. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values. If either the Baseline or post-randomization value was missing, the change from Baseline is set to missing as well. If measurements were taken in triplicate, then the mean of the triplicate measurements was used as the Baseline. AUC with respect to that time interval was calculated using the linear trapezoidal rule. The weighted mean was determined by dividing the AUC by the observed length of the collection interval (time of last assessment - time of first assessment in hours). In order for the AUC to be calculated, the first and last time points and at least one additional assessment falling between the two must be non-missing.
Time Frame: Baseline and at pre-breakfast on Days -1 and 14, and then at 0.5, 1, 1.5, 2 and 3 hours post dose.
Population: PD Population
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 14 | 13 | 12 | 14 | 12
pmol/L
  Weighted mean (0-12), Day 7 | 6.146 [-12.944 to 25.236] | -19.241 [-39.283 to 0.801] | -47.290 [-89.816 to -4.764] | -36.334 [-67.090 to -5.578] | 5.979 [-20.154 to 32.112]
  Weighted mean (0-12), Day 14 | 21.751 [4.762 to 38.739] | 6.672 [-15.624 to 28.968] | -42.657 [-91.850 to 6.535] | -33.753 [-61.363 to -6.143] | 17.328 [-4.094 to 38.750]
  Weighted mean (0-24), Day 14 | 22.127 [5.128 to 39.127] | 4.626 [-15.718 to 24.970] | -35.220 [-70.650 to 0.209] | -31.067 [-65.498 to 3.363] | 18.848 [-2.177 to 39.874]
Statistical Analysis 1: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = -28.619, 95% CI 2-sided [-59.25 to 2.01]
Statistical Analysis 2: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = -47.898, 95% CI 2-sided [-79.23 to -16.56]
Statistical Analysis 3: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = -24.665, 95% CI 2-sided [-55.53 to 6.20]
Statistical Analysis 4: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = -5.438, 95% CI 2-sided [-36.76 to 25.89]
Statistical Analysis 5: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = -23.181, 95% CI 2-sided [-55.00 to 8.63]
Statistical Analysis 6: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = -42.460, 95% CI 2-sided [-75.18 to -9.74]
Statistical Analysis 7: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 7; Test type: Superiority or Other; Mean Difference (Net) = -19.227, 95% CI 2-sided [-51.83 to 13.37]
Statistical Analysis 8: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -18.435, 95% CI 2-sided [-49.15 to 12.28]
Statistical Analysis 9: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -58.658, 95% CI 2-sided [-90.08 to -27.24]
Statistical Analysis 10: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -37.006, 95% CI 2-sided [-67.96 to -6.05]
Statistical Analysis 11: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -9.896, 95% CI 2-sided [-41.31 to 21.52]
Statistical Analysis 12: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -8.539, 95% CI 2-sided [-40.44 to 23.36]
Statistical Analysis 13: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -48.762, 95% CI 2-sided [-81.58 to -15.95]
Statistical Analysis 14: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Weighted Mean (0-12), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -27.110, 95% CI 2-sided [-59.80 to 5.58]
Statistical Analysis 15: Comparison: Placebo vs GSK1292263 75 mg; Placebo vs GSK1292263 75 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -20.359, 95% CI 2-sided [-48.95 to 8.23]
Statistical Analysis 16: Comparison: Placebo vs GSK1292263 300 mg; Placebo vs GSK1292263 300 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -53.712, 95% CI 2-sided [-82.92 to -24.50]
Statistical Analysis 17: Comparison: Placebo vs GSK1292263 600 mg; Placebo vs GSK1292263 600 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -37.552, 95% CI 2-sided [-66.24 to -8.86]
Statistical Analysis 18: Comparison: Placebo vs Sitagliptin 50 mg; Placebo vs Sitagliptin 50 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -7.963, 95% CI 2-sided [-37.20 to 21.27]
Statistical Analysis 19: Comparison: GSK1292263 75 mg vs Sitagliptin 50 mg; GSK1292263 75 mg vs Sitagliptin 50 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -12.397, 95% CI 2-sided [-42.10 to 17.30]
Statistical Analysis 20: Comparison: GSK1292263 300 mg vs Sitagliptin 50 mg; GSK1292263 300 mg vs Sitagliptin 50 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -45.749, 95% CI 2-sided [-76.20 to -15.30]
Statistical Analysis 21: Comparison: GSK1292263 600 mg vs Sitagliptin 50 mg; GSK1292263 600 mg vs Sitagliptin 50 mg: Weighted Mean (0-24), Day 14; Test type: Superiority or Other; Mean Difference (Net) = -29.590, 95% CI 2-sided [-59.82 to 0.64]

39. Primary Outcome: Number of Participants With Relationship Between GSK1292263 Drug Exposures and Pharmacodynamic Parameters (Part B)
Description: Data was not collected for this outcome measure.
Time Frame: At pre-breakfast on Days -1 and 14, and then at 0.5, 1, 1.5, 2 and 3 hours post dose
Population: PD Population. No data was collected for this outcome measure.
Arm/Group | Placebo | GSK1292263 75 mg | GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were reported up to 10 days after discharge (Day 2) in Part A and up to 10 days after discharge (Day 15 ) in Part B.
Description: AEs and SAEs were reported for the Safety Population which consisted of all participants enrolled in the study and who had received at least one dose of study drug.
Groups:
- Part A - GSK1292263 300 mg: Participants received a single dose of oral 300 mg tablet of GSK1292263 on Day 1 immediately after eating the breakfast meal. Participants also received their usual metformin monotherapy (>=1000 mg per day).
- Part B - Placebo: Participants received 3 tablets of matching placebo BID along with metformin for 14 days.
- Part B - GSK1292263 75 mg: Participant received 1 tablet of 75 mg of GSK1292263 and 2 tablets of matching placebo along with metformin BID for 14 days.
- Part B - GSK1292263 300 mg: Participant received 1 tablet of 200 mg, 1 tablet of 75 mg and 1 tablet of 25 mg (all GSK1292263) along with metformin BID for 14 days.
Arm/Group | Part A - GSK1292263 300 mg | Part B - Placebo | Part B - GSK1292263 75 mg | Part B - GSK1292263 300 mg | GSK1292263 600 mg | Sitagliptin 50 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/14 | 0/13 | 0/12 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/14 | 0/13 | 0/12 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/6 | 2/14 | 3/13 | 3/12 | 4/15 | 5/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - GSK1292263 300 mg (N=6) | Part B - Placebo (N=14) | Part B - GSK1292263 75 mg (N=13) | Part B - GSK1292263 300 mg (N=12) | GSK1292263 600 mg (N=15) | Sitagliptin 50 mg (N=13)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Infected sebaceous cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.